CLINICAL TRIAL: NCT00536484
Title: A 12-Week, Randomized, Double-Blind, Placebo-Controlled, Parallel-Group, Multicenter Trial To Evaluate The Efficacy And Safety Of A Fesoterodine Flexible Dose Regimen In Patients With Overactive Bladder.
Brief Title: Fesoterodine Flexible Dose Study
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Director, Clinical Trial Disclosure Group, Pfizer Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A0221014
Record Dates: First submitted 2007-09-25; First posted 2007-09-27 (Estimated); Results first posted 2009-09-11 (Estimated); Last update posted 2009-09-15 (Estimated); Status verified 2009-09

CONDITIONS: Overactive Bladder
Keywords: Overactive Bladder
MeSH Terms: conditions — Urinary Bladder, Overactive | interventions — fesoterodine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fesoterodine (Double-Blind) (Experimental)
  Interventions: Drug: Fesoterodine
- Placebo (Double-Blind) (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Fesoterodine — 4mg tablets once daily for 2 weeks, then either 4mg or 8mg tablets once daily for 10 weeks. Subjects were instructed to take 1 tablet every evening within 4 hours prior to bedtime with water, swallowed whole without chewing.
  Arms: Fesoterodine (Double-Blind)
Drug: Placebo — Matched placebo tablets once daily for 12 weeks. Subjects were instructed to take 1 tablet every evening within 4 hours prior to bedtime with water, swallowed whole without chewing.
  Arms: Placebo (Double-Blind)

SUMMARY:
This Phase 3B study is designed to test if a fesoterodine flexible dose regimen is more effective than placebo in reducing micturition frequency and other overactive bladder (OAB) symptoms, e.g., urgency, urgency incontinence episodes in patients with overactive bladder and if the fesoterodine regimen is safe and well tolerated.

ELIGIBILITY:
Inclusion Criteria:

* Overactive bladder symptoms for greater than or equal to 3 months.
* Mean urinary frequency of greater than or equal to 8 micturitions per 24 hours in bladder diary.
* Mean number of Urgency episodes greater than or equal to 3 per 24 hours in bladder diary.

Exclusion Criteria:

* Contraindication to fesoterodine (antimuscarinics).
* Known etiology of OAB (e.g., neurogenic, local urinary tract pathology).
* Previous history of acute urinary retention requiring catheterization or severe voiding difficulties in the judgment of the investigator, prior to baseline.
* Unable to follow the study procedures, including completion of self-administered bladder diary and patient reported outcome questionnaires.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 896 (Actual)
Dates: Start 2007-08; Primary Completion 2008-03 (Actual); Study Completion 2008-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (84):
- United States (84):
  - Pfizer Investigational Site, Mobile, Alabama
  - Pfizer Investigational Site, Chandler, Arizona
  - Pfizer Investigational Site, Peoria, Arizona
  - Pfizer Investigational Site, Tucson, Arizona
  - Pfizer Investigational Site, Rancho Cordova, California
  - Pfizer Investigational Site, Sacramento, California
  - Pfizer Investigational Site, San Diego, California
  - Pfizer Investigational Site, Denver, Colorado
  - Pfizer Investigational Site, Englewood, Colorado
  - Pfizer Investigational Site, New Britain, Connecticut
  - Pfizer Investigational Site, Aventura, Florida
  - Pfizer Investigational Site, Bonita Springs, Florida
  - Pfizer Investigational Site, Hollywood, Florida
  - Pfizer Investigational Site, Lake Worth, Florida
  - Pfizer Investigational Site, Miami, Florida
  - Pfizer Investigational Site, Naples, Florida
  - Pfizer Investigational Site, Pembroke Pines, Florida
  - Pfizer Investigational Site, St. Petersburg, Florida
  - Pfizer Investigational Site, Stuart, Florida
  - Pfizer Investigational Site, Tallahassee, Florida
  - Pfizer Investigational Site, Chicago, Illinois
  - Pfizer Investigational Site, Evansville, Indiana
  - Pfizer Investigational Site, Jeffersonville, Indiana
  - Pfizer Investigational Site, Newburgh, Indiana
  - Pfizer Investigational Site, Iowa City, Iowa
  - Pfizer Investigational Site, Overland Park, Kansas
  - Pfizer Investigational Site, Pratt, Kansas
  - Pfizer Investigational Site, Lexington, Kentucky
  - Pfizer Investigational Site, Louisville, Kentucky
  - Pfizer Investigational Site, Madisonville, Kentucky
  - Pfizer Investigational Site, Baltimore, Maryland
  - Pfizer Investigational Site, Bel Air, Maryland
  - Pfizer Investigational Site, Milford, Massachusetts
  - Pfizer Investigational Site, Springfield, Massachusetts
  - Pfizer Investigational Site, West Yarmouth, Massachusetts
  - Pfizer Investigational Site, Ann Arbor, Michigan
  - Pfizer Investigational Site, Paw Paw, Michigan
  - Pfizer Investigational Site, Royal Oak, Michigan
  - Pfizer Investigational Site, Troy, Michigan
  - Pfizer Investigational Site, Picayune, Mississippi
  - Pfizer Investigational Site, St Louis, Missouri
  - Pfizer Investigational Site, Lincoln, Nebraska
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Las Vegas, Nevada
  - Pfizer Investigational Site, New Brunswick, New Jersey
  - Pfizer Investigational Site, Garden City, New York
  - Pfizer Investigational Site, Kingston, New York
  - Pfizer Investigational Site, Manlius, New York
  - Pfizer Investigational Site, New York, New York
  - Pfizer Investigational Site, Poughkeepsie, New York
  - Pfizer Investigational Site, Rochester, New York
  - Pfizer Investigational Site, Syracuse, New York
  - Pfizer Investigational Site, Williamsville, New York
  - Pfizer Investigational Site, Cary, North Carolina
  - Pfizer Investigational Site, Charlotte, North Carolina
  - Pfizer Investigational Site, Raleigh, North Carolina
  - Pfizer Investigational Site, Winston-Salem, North Carolina
  - Pfizer Investigational Site, Cincinnati, Ohio
  - Pfizer Investigational Site, Bethany, Oklahoma
  - Pfizer Investigational Site, Norman, Oklahoma
  - Pfizer Investigational Site, Portland, Oregon
  - Pfizer Investigational Site, Lansdale, Pennsylvania
  - Pfizer Investigational Site, Philadelphia, Pennsylvania
  - Pfizer Investigational Site, Sellersville, Pennsylvania
  - Pfizer Investigational Site, State College, Pennsylvania
  - Pfizer Investigational Site, Cranston, Rhode Island
  - Pfizer Investigational Site, Cumberland, Rhode Island
  - Pfizer Investigational Site, Warwick, Rhode Island
  - Pfizer Investigational Site, Mt. Pleasant, South Carolina
  - Pfizer Investigational Site, Bristol, Tennessee
  - Pfizer Investigational Site, Johnson City, Tennessee
  - Pfizer Investigational Site, Nashville, Tennessee
  - Pfizer Investigational Site, New Tazewell, Tennessee
  - Pfizer Investigational Site, Bryan, Texas
  - Pfizer Investigational Site, Corpus Christi, Texas
  - Pfizer Investigational Site, Dallas, Texas
  - Pfizer Investigational Site, Houston, Texas
  - Pfizer Investigational Site, Longview, Texas
  - Pfizer Investigational Site, San Antonio, Texas
  - Pfizer Investigational Site, Arlington, Virginia
  - Pfizer Investigational Site, Norfolk, Virginia
  - Pfizer Investigational Site, Richmond, Virginia
  - Pfizer Investigational Site, Mountlake Terrace, Washington
  - Pfizer Investigational Site, Spokane, Washington

REFERENCES:
- [Derived] Stoniute A, Madhuvrata P, Still M, Barron-Millar E, Nabi G, Omar MI. Oral anticholinergic drugs versus placebo or no treatment for managing overactive bladder syndrome in adults. Cochrane Database Syst Rev. 2023 May 9;5(5):CD003781. doi: 10.1002/14651858.CD003781.pub3. PMID 37160401
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A0221014&StudyName=Fesoterodine%20flexible%20dose%20study

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were screened at 90 centers in the United States; in 88 centers, participants were randomized.
Pre-assignment Details: The study consisted of a 2-week no-treatment screening period and a 12-week double-blind treatment period. Participants with bothersome overactive bladder (OAB) symptoms who met all entry criteria at baseline (end of screening) were randomized.
Groups:
- Placebo: All randomized participants were treated with placebo once daily for the first 2 weeks of treatment. The dose remained as placebo once daily or changed to matching placebo (for 8 mg) once daily for the next 10 weeks based on discussion between investigator and participant.
- Fesoterodine: All randomized participants were treated with fesoterodine 4mg once daily for the first 2 weeks of treatment. The dose remained at 4 mg once daily or increased to 8 mg once daily for the next 10 weeks based on discussion between investigator and participant.
Period: Overall Study
Arm/Group | Placebo | Fesoterodine
Started | 445 (448 participants randomised; 3 not treated) | 438 (448 participants randomised; 10 not treated)
Completed | 385 (88 completed on matched 4mg dose and 297 on matched 8mg dose) | 382 (134 completed on 4mg dose and 248 on 8mg dose)
Not Completed | 60 | 56
Not completed — Adverse Event | 21 | 34
Not completed — Withdrawal by Subject | 11 | 11
Not completed — Lost to Follow-up | 8 | 6
Not completed — Lack of Efficacy | 16 | 5
Not completed — Other | 4 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo | Fesoterodine | Total
Number analyzed (Participants) | 445 | 438 | 883
Age Continuous [Mean (Standard Deviation); unit: years] | 60.1 (12.9) | 59.7 (13.7) | 59.9 (13.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 368 | 364 | 732.0
  Male | 77 | 74 | 151.0

OUTCOME MEASURES:

1. Primary Outcome: Change in Mean Number of Micturition Episodes Per 24 Hours at Week 12 Relative to Baseline.
Description: The number of micturitions per 24 hours was calculated as the sum of all micturitions divided by the total number of diary days collected at that visit.
  Change: mean at Week 12 minus mean at Baseline
Time Frame: Baseline and Week 12
Population: Participants in the Full Analysis Set (FAS) with non-missing numerical change from baseline to Week 12 (last observation carried forward [LOCF)). The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 valid efficacy assessment, either at baseline or post baseline.
Measure: Least Squares Mean (Standard Error); unit: number of episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 434 | 428
number of episodes per 24 hours | -2.1 (0.1) | -2.9 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Null hypothesis: the mean change from baseline in micturitions per 24 hours in the fesoterodine group is the same as in the placebo group at Week 12. A sample size of 350 in each arm had at least 85% power to detect a difference of 0.8 between flexible dose fesoterodine & placebo assuming a standard deviation of 3.52 using a 2-sample t-test with a 0.05 2-sided significance level. Accounting for 10% of randomized subjects not having the primary endpoint data, 390 subjects were needed in each arm; Test type: Superiority or Other; p = 0.0002, ANCOVA — Significance level p <0.05; Terms for treatment, center and baseline as covariate and baseline by treatment interaction; Mean Difference (Final Values) = -0.7, 95% CI [-1.1 to -0.4], Standard Error of Mean 0.2 — The LS mean difference & 95% CI were calculated at mean baseline = 12.9 (centered baseline used in model)

2. Secondary Outcome: Change in Mean Number of Micturition Episodes Per 24 Hours Relative to Baseline
Description: The number of micturitions per 24 hours was calculated as the sum of all micturitions divided by the total number of diary days collected at that visit.
  Change: mean at observation minus mean at baseline
Time Frame: Baseline, Week 2 and Week 6
Population: Participants in the Full Analysis Set (FAS) with non-missing numerical change from baseline to Week 2 or Week 6 (last observation carried forward [LOCF]).
  The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 valid efficacy assessment, either at baseline or post baseline (n=placebo; n=fesoterodine)
Measure: Least Squares Mean (Standard Error); unit: number of episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 435
number of episodes per 24 hours
  Week 2 (n=431; n=427) | -1.3 (0.1) | -1.8 (0.1)
  Week 6 (n=434; n=428) | -2.0 (0.1) | -2.7 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 2 minus Baseline; Test type: Superiority or Other; p = 0.0136, ANCOVA — Significance level p <0.05; Terms for center, treatment, baseline covariate and baseline by treatment interaction; Mean Difference (Final Values) = -0.4, 95% CI [-0.8 to -0.1], Standard Error of Mean 0.2 — Since centered baseline was used in the model, the LS mean difference and its 95% CI were calculated at mean baseline
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Week 6 minus Baseline; Test type: Superiority or Other; p = 0.0002, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline as covariate and baseline by treatment interaction; Mean Difference (Final Values) = -0.7, 95% CI [-1.1 to -0.3], Standard Error of Mean 0.2 — Since centered baseline was used in the model, the LS mean difference and its 95% CI were calculated at mean baseline

3. Secondary Outcome: Change in Number of Urgency Episodes Per 24 Hours Relative to Baseline
Description: Change in number of urgency episodes (urinary sensation scale [USS] rating of 3 or more) recorded in the bladder diary. Scale: 0=no feeling of urgency to 5=unable to hold; leak urine. The number of urgency episodes per 24 hours was calculated as the sum of all urgency episodes divided by the total number of diary days collected at that visit.
Time Frame: Baseline, Week 2, Week 6 and Week 12
Population: Number of subjects with Baseline Urgency Episodes >0 per 24 hours and non missing change from baseline to Week 2, Week 6 (last observation carried forward [LOCF]) or Week 12 (LOCF). Only subjects with at least 1 episode during baseline 3-day diary period were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: number of episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 444 | 437
number of episodes per 24 hours
  Week 2 (n=431; n=427) | -1.9 (0.2) | -2.3 (0.2)
  Week 6 (n=434; n=428) | -2.9 (0.2) | -3.5 (0.2)
  Week 12 (n=434; n=428) | -3.0 (0.2) | -4.0 (0.2)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 2 minus Baseline; Test type: Superiority or Other; p = 0.1057, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -0.4, 95% CI [-0.9 to 0.1], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Week 6 minus Baseline; Test type: Superiority or Other; p = 0.0338, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -0.6, 95% CI [-1.1 to -0.0], Standard Error of Mean 0.3
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline; Test type: Superiority or Other; p = 0.0003, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -1.0, 95% CI [-1.5 to -0.5], Standard Error of Mean 0.3

4. Secondary Outcome: Change in Number of Severe Urgency Episodes Per 24 Hours Relative to Baseline
Description: Change in number of severe urgency episodes (urinary sensation scale [USS] rating of 4 or more) recorded in the bladder diary. Scale: 0=no feeling of urgency to 5=unable to hold; leak urine. Number of severe urgency episodes per 24 hours calculated as sum of all severe urgency episodes divided by total number of diary days collected at that visit.
Time Frame: Baseline, Week 2, Week 6 and Week 12
Population: Number of subjects with baseline severe urgency episodes >0 per 24 hours and non-missing change from baseline to Week 2, Week 6 (last observation carried forward [LOCF]) or Week 12 (LOCF). Only those with at least 1 episode during baseline 3-day diary period were included.
Measure: Least Squares Mean (Standard Error); unit: number of episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 405 | 412
number of episodes per 24 hours
  Week 2 (n=393; n=403) | -1.6 (0.1) | -1.8 (0.1)
  Week 6 (n=396; n=404) | -2.2 (0.1) | -2.6 (0.1)
  Week 12 (n=396; n=404) | -2.2 (0.1) | -2.9 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 2 minus Baseline; Test type: Superiority or Other; p = 0.1666, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -0.3, 95% CI [-0.6 to 0.1], Standard Error of Mean 0.2
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Week 6 minus Baseline; Test type: Superiority or Other; p = 0.0506, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -0.4, 95% CI [-0.8 to 0.0], Standard Error of Mean 0.2
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline; Test type: Superiority or Other; p = 0.0014, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -0.6, 95% CI [-1.0 to -0.2], Standard Error of Mean 0.2

5. Secondary Outcome: Change in Number of Urgency Urinary Incontinence (UUI) Episodes Per 24 Hours Relative to Baseline
Description: Change in number of UUI episodes (urinary sensation scale [USS] rating of 5) recorded in the bladder diary. Scale: 0=no feeling of urgency to 5=unable to hold; leak urine
Time Frame: Baseline, Week 2, Week 6 and Week 12
Population: Number of subjects with Baseline UUI >0 per 24 hours and non-missing change from baseline to Week 2, Week 6 (last observation carried forward [LOCF]) or Week 12 (LOCF). Only subjects with at least 1 episode during baseline 3-day diary period were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: number of episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 260 | 257
number of episodes per 24 hours
  Week 2 (n=255; n=251) | -0.9 (0.1) | -1.1 (0.1)
  Week 6 (n=257; n=251) | -1.2 (0.1) | -1.5 (0.1)
  week 12 (n=257; n=251) | -1.2 (0.1) | -1.5 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 2 minus Baseline; Test type: Superiority or Other; p = 0.2054, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline as covariate and baseline by treatment interaction; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to 0.1], Standard Error of Mean 0.1 — Since centered baseline was used in the model, the LS mean difference and its 95% CI were calculated at mean baseline
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Week 6 minus Baseline; Test type: Superiority or Other; p = 0.0225, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline as covariate and baseline by treatment interaction; Mean Difference (Final Values) = -0.3, 95% CI [-0.6 to -0.0], Standard Error of Mean 0.1 — Since centered baseline was used in the model, the LS mean difference and its 95% CI were calculated at mean baseline
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline; Test type: Superiority or Other; p = 0.0167, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline as covariate and baseline by treatment interaction; Mean Difference (Final Values) = -0.3, 95% CI [-0.6 to -0.1], Standard Error of Mean 0.1 — Since centered baseline was used in the model, the LS mean difference and its 95% CI were calculated at mean baseline

6. Secondary Outcome: Change in Nocturnal Micturition Episodes Per 24 Hours Relative to Baseline
Description: Change in number of nocturnal micturitions (NM) recorded in the bladder diary. NM were defined as micturitions that occurred between the time the subject went to bed and the time he or she arose to start the next day. The number of NM per 24 hours was calculated as the sum of all NM divided by the total number of diary days collected at that visit.
Time Frame: Baseline, Week 2, Week 6 and Week 12
Population: Number of subjects with Baseline Nocturnal Micturitions >0 per 24 and non-missing change from baseline to Week 2, Week 6 (last observation carried forward [LOCF]) or Week 12 (LOCF). Only subjects with at least 1 episode during baseline 3-day diary period were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: number of episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 433 | 427
number of episodes per 24 hours
  Week 2 (n=420; n=417) | -0.5 (0.1) | -0.5 (0.1)
  Week 6 (n=423; n=418) | -0.7 (0.1) | -0.7 (0.1)
  Week 12 (n=423; n=418) | -0.7 (0.1) | -0.8 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 2 minus Baseline; Test type: Superiority or Other; p = 0.8019, ANOVA — Significance level p <0.05; Mean Difference (Final Values) = -0.0, 95% CI [-0.2 to 0.1], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Week 6 minus Baseline; Test type: Superiority or Other; p = 0.3881, ANOVA — Significance level p <0.05; Mean Difference (Final Values) = -0.1, 95% CI [-0.2 to 0.1], Standard Error of Mean 0.1
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline; Test type: Superiority or Other; p = 0.3240, ANOVA — Significance level p <0.05; Mean Difference (Final Values) = -0.1, 95% CI [-0.2 to 0.1], Standard Error of Mean 0.1

7. Secondary Outcome: Change in Number of Nocturnal Urgency Episodes Per 24 Hours Relative to Baseline
Description: Change in number of nocturnal urgency episodes (NUE) recorded in bladder diary. NUE had urinary sensation scale (USS) rating of 3 or more that occurred between time subject went to bed and time he or she arose to start next day. Number of NUE per 24 hours was calculated as sum of all NUE divided by total number of diary days collected at that visit
Time Frame: Baseline, Week 2, Week 6 and Week 12
Population: Number of subjects with Nocturnal Urgency Episodes >0 per 24 hours and non-missing change from baseline to Week 2, Week 6 (last observation carried forward [LOCF]) or Week 12 (LOCF). Only subjects with at least 1 episode during baseline 3-day diary period were included in analysis.
Measure: Least Squares Mean (Standard Error); unit: number of episodes per 24 hours
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 424 | 418
number of episodes per 24 hours
  Week 2 (n=411; n=408) | -0.6 (0.1) | -0.6 (0.1)
  Week 6 (n=414; n=409) | -0.8 (0.1) | -0.9 (0.1)
  Week 12 (n=414; n=409) | -0.9 (0.1) | -1.0 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 2 minus Baseline; Test type: Superiority or Other; p = 0.8279, ANOVA — Significance level p <0.05; Mean Difference (Final Values) = -0.0, 95% CI [-0.2 to 0.1], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Week 6 minus Baseline; Test type: Superiority or Other; p = 0.5059, ANOVA — Significance level p <0.05; Mean Difference (Final Values) = -0.1, 95% CI [-0.2 to 0.1], Standard Error of Mean 0.1
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline; Test type: Superiority or Other; p = 0.0806, ANOVA — Significance level p <0.05; Mean Difference (Final Values) = -0.2, 95% CI [-0.4 to 0.0], Standard Error of Mean 0.1

8. Secondary Outcome: Change in Frequency-urgency Sum Per 24 Hours Relative to Baseline
Description: Change in frequency urgency sum is total urinary sensation scale (USS) ratings recorded for all micturitions in 24-hour day. Number of USS ratings per 24 hours is sum of all USS ratings divided by the total diary days collected at that visit. USS scale: 1=No feeling of urgency to 5=Unable to hold:leak urine. Numerical decrease indicates improvement
Time Frame: Baseline, Week 2, Week 6 and Week 12
Population: Participants in the Full Analysis Set (FAS) with non-missing numerical change from baseline to Week 2, Week 6 or Week 12 (last observation carried forward [LOCF]).
  Number analyzed=participants at Week 12 LOCF.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 435
scores on a scale
  Week 2 (n=431; n=427) | -6.5 (0.5) | -8.3 (0.5)
  Week 6 (n=434; n=428) | -9.8 (0.6) | -12.5 (0.6)
  Week 12 (n=434; n=428) | -10.3 (0.6) | -13.6 (0.6)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 2 minus Baseline; Test type: Superiority or Other; p = 0.0203, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -1.7, 95% CI [-3.2 to -0.3], Standard Error of Mean 0.7
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Week 6 minus Baseline; Test type: Superiority or Other; p = 0.0007, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -2.7, 95% CI [-4.2 to -1.1], Standard Error of Mean 0.8
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -3.3, 95% CI [-4.9 to -1.7], Standard Error of Mean 0.8

9. Secondary Outcome: Change in Overactive Bladder Questionnaire (OAB-q) at Week 12 Relative to Baseline - Symptom Bother Scale
Description: Each item rated by subject on a Likert scale 1 (least symptom bother) to 6 (most symptom bother). Raw scores were transformed to a score from 0 to 100. Once transformed a negative change indicates improvement.
  Change: mean at Week 12 minus mean at baseline
Time Frame: Baseline and Week 12
Population: Participants in the Full Analysis Set (FAS) with non-missing numerical change from baseline to Week 12.
  The FAS included all participants who took at least 1 dose of assigned study drug and had at least 1 valid efficacy assessment, either at baseline or post baseline
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 384 | 378
scores on a scale | -20.0 (1.1) | -27.8 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline as covariate and baseline by treatment interaction; Mean Difference (Final Values) = -7.8, 95% CI [-10.7 to -4.9], Standard Error of Mean 1.5 — Since centered baseline was used in the model, the LS mean difference and its 95% CI were calculated at mean baseline

10. Secondary Outcome: Change in Overactive Bladder Questionnaire (OAB-q) at Week 12 Relative to Baseline - Health Related Quality of Life (HRQL) Subscales
Description: Each item rated by subject on a Likert scale 1 (least symptom bother) to 6 (most symptom bother). Raw scores were transformed to a score from 0 to 100. Once transformed a positive change indicates improvement.
  Change: mean at Week 12 minus mean at baseline.
Time Frame: Baseline and Week 12
Population: as for outcome 9
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 435
scores on a scale
  HRQL concern domain (n=383; n=372) | 20.9 (1.1) | 29.3 (1.2)
  HRQL coping domain (n=383; n=372) | 20.2 (1.2) | 27.2 (1.2)
  HRQL sleep domain (n=383; n=372) | 21.2 (1.2) | 25.9 (1.2)
  HRQL social interaction domain (n=380; n=372) | 11.6 (0.8) | 15.3 (0.8)
  HRQL scale score total (n=380; n=372) | 18.9 (1.0) | 25.1 (1.0)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline Concern domain; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline as covariate and baseline by treatment interaction; Mean Difference (Final Values) = 8.4, 95% CI [5.3 to 11.5], Standard Error of Mean 1.6 — Since centered baseline was used in the model, the LS mean difference and its 95% CI were calculated at mean baseline
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline Coping domain; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline as covariate and baseline by treatment interaction; Mean Difference (Final Values) = 7.1, 95% CI [3.9 to 10.2], Standard Error of Mean 1.6 — Since centered baseline was used in the model, the LS mean difference and its 95% CI were calculated at mean baseline
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline Sleep domain; Test type: Superiority or Other; p = 0.0036, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline as covariate; Mean Difference (Final Values) = 4.7, 95% CI [1.5 to 7.8], Standard Error of Mean 1.6
Statistical Analysis 4: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline Social interaction domain; Test type: Superiority or Other; p = 0.0007, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline as covariate and baseline by treatment interaction; Mean Difference (Final Values) = 3.7, 95% CI [1.6 to 5.8], Standard Error of Mean 1.1 — Since centered baseline was used in the model, the LS mean difference and its 95% CI were calculated at mean baseline
Statistical Analysis 5: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline HRQL scale score total; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline as covariate and baseline by treatment interaction; Mean Difference (Final Values) = 6.2, 95% CI [3.6 to 8.9], Standard Error of Mean 1.3 — Since centered baseline was used in the model, the LS mean difference and its 95% CI were calculated at mean baseline

11. Secondary Outcome: Categorical Change in Patient Perception of Bladder Condition (PPBC) Score Relative to Baseline
Description: PPBC scale range: 1='does not cause me any problems at all' to 6='causes me many severe problems'. Major improvement=negative score change of 2 or more from baseline; minor improvement=negative score change of 1 or more from baseline; no change=0 score change from baseline; Deterioration=positive score change from baseline
Time Frame: Baseline, Week 2, Week 6 and Week 12
Population: Participants in the Full Analysis Set (FAS) with non-missing baseline values and Week 2, Week 6 (last observation carried forward [LOCF]) or Week 12 (LOCF) values.
  Number analyzed=participants at Week 12 LOCF.
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 435
percentage of participants
  Week 2 (n=440; n=434): major improvement | 13.2 | 16.6
  Week 2: minor improvement | 34.8 | 39.4
  Week 2: no change | 45.2 | 39.4
  Week 2: deterioration | 6.8 | 4.6
  Week 6 (n=442; n=435): major improvement | 24.7 | 32.4
  Week 6: minor improvement | 34.8 | 35.9
  Week 6: no change | 33.5 | 27.8
  Week 6: deterioration | 7.0 | 3.9
  Week 12 (n=442; n=435): major improvement | 29.2 | 36.8
  Week 12: minor improvement | 31.0 | 34.5
  Week 12: no change | 33.0 | 25.5
  Week 12: deterioration | 6.8 | 3.2
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference at Week 2; Test type: Superiority or Other; p = 0.0087, Cochran-Mantel-Haenszel — Significance level p <0.05; The CMH test used modified ridit scores which were based on the ranks of the observations rather than the observed values
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Treatment difference at Week 6; Test type: Superiority or Other; p = 0.0008, Cochran-Mantel-Haenszel — Significance level p <0.05; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Treatment difference at Week 12; Test type: Superiority or Other; p = 0.0006, Cochran-Mantel-Haenszel — Significance level p <0.05; [statistical method as in outcome 11, analysis 1]

12. Secondary Outcome: Categorical Change in Urgency Perception Scale (UPS) Relative to Baseline
Description: UPS scores range from 0 ("I am usually not able to hold urine") to 2 ("I am usually able to finish what I am doing before going to the toilet [without leaking]"). Improvement: positive score change; No change: score change=0; Deterioration: negative score change
Time Frame: Baseline, Week 2, Week 6 and Week 12
Population: as for outcome 11
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 435
percentage of participants
  Week 2 (n=441; n=434): improvement | 22.9 | 29.3
  Week 2: no change | 69.2 | 64.5
  Week 2: deterioration | 7.9 | 6.2
  Week 6 (n=443; n=435): improvement | 30.2 | 37.5
  Week 6: no change | 65.0 | 58.6
  Week 6: deterioration | 4.7 | 3.9
  Week 12 (n=443; n=435): improvement | 30.9 | 41.8
  Week 12: no change | 62.3 | 52.4
  Week 12: deterioration | 6.8 | 5.7
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Treatment difference at Week 2; Test type: Superiority or Other; p = 0.0129, Cochran-Mantel-Haenszel — Significance level p <0.05; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Treatment difference at Week 6; Test type: Superiority or Other; p = 0.0100, Cochran-Mantel-Haenszel — Significance level p <0.05; [statistical method as in outcome 11, analysis 1]
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Treatment difference at Week 12; Test type: Superiority or Other; p = 0.0009, Cochran-Mantel-Haenszel — Significance level p <0.05; [statistical method as in outcome 11, analysis 1]

13. Secondary Outcome: Change in Urgency Severity Visual Analog Scale (VAS) Relative to Baseline
Description: The urgency severity VAS Scale records the subject's assessment of the severity of urgency. VAS scale ranges from 1 'Very Mild' to 10 'Very Severe'. Negative change indicated improvement.
  Change: mean at observation minus mean at baseline.
Time Frame: Baseline, Week 2, Week 6 and Week 12
Population: as for outcome 8
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | Placebo | Fesoterodine
Number analyzed (Participants) | 445 | 435
scores on a scale
  Week 2 (n=441; n=432) | -0.8 (0.1) | -1.4 (0.1)
  Week 6 (n=443; n=434) | -1.4 (0.1) | -2.2 (0.1)
  Week 12 (n=443; n=434) | -1.4 (0.1) | -2.4 (0.1)
Statistical Analysis 1: Comparison: Placebo vs Fesoterodine; Week 2 minus Baseline; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -0.6, 95% CI [-0.9 to -0.4], Standard Error of Mean 0.1
Statistical Analysis 2: Comparison: Placebo vs Fesoterodine; Week 6 minus Baseline; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -0.8, 95% CI [-1.1 to -0.5], Standard Error of Mean 0.1
Statistical Analysis 3: Comparison: Placebo vs Fesoterodine; Week 12 minus Baseline; Test type: Superiority or Other; p < 0.0001, ANCOVA — Significance level p <0.05; Terms for center, treatment and baseline covariate; Mean Difference (Final Values) = -1.0, 95% CI [-1.3 to -0.7], Standard Error of Mean 0.2

ADVERSE EVENTS:
Arm/Group | Placebo | Fesoterodine
Serious Adverse Events (participants affected / at risk) | 7 | 5
Other Adverse Events (participants affected / at risk) | 130 | 199
SERIOUS ADVERSE EVENTS; cells are participants affected / at risk:
Term (organ system) | Placebo | Fesoterodine
Intestinal obstruction (Gastrointestinal disorders) | 0/445 | 1/438
Nausea (Gastrointestinal disorders) | 1/445 | 0/438
Vomiting (Gastrointestinal disorders) | 1/445 | 0/438
Chest pain (General disorders) | 1/445 | 0/438
Cellulitis (Infections and infestations) | 1/445 | 0/438
Pneumonia (Infections and infestations) | 2/445 | 2/438
Urinary tract infection (Infections and infestations) | 2/445 | 0/438
Fall (Injury, poisoning and procedural complications) | 1/445 | 0/438
Arthralgia (Musculoskeletal and connective tissue disorders) | 1/445 | 0/438
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0/445 | 1/438
Asthma (Respiratory, thoracic and mediastinal disorders) | 0/445 | 1/438
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 1/445 | 0/438
Deep vein thrombosis (Vascular disorders) | 0/445 | 1/438
Dehydration (Metabolism and nutrition disorders) | 1/445 | 0/438
Hypotension (Vascular disorders) | 1/445 | 0/438
Staphylococcal sepsis (Infections and infestations) | 0/445 | 1/438
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected / at risk:
Term (organ system) | Placebo | Fesoterodine
Dry eye (Eye disorders) | 8/445 | 13/438
Constipation (Gastrointestinal disorders) | 25/445 | 48/438
Diarrhoea (Gastrointestinal disorders) | 19/445 | 9/438
Dry mouth (Gastrointestinal disorders) | 34/445 | 113/438
Nausea (Gastrointestinal disorders) | 18/445 | 6/438
Fatigue (General disorders) | 2/445 | 11/438
Nasopharyngitis (Infections and infestations) | 25/445 | 19/438
Upper respiratory tract infection (Infections and infestations) | 23/445 | 21/438
Urinary tract infection (Infections and infestations) | 12/445 | 8/438
Headache (Nervous system disorders) | 15/445 | 19/438
Insomnia (Psychiatric disorders) | 2/445 | 11/438
Cough (Respiratory, thoracic and mediastinal disorders) | 2/445 | 9/438
Dry throat (Respiratory, thoracic and mediastinal disorders) | 1/445 | 9/438

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of < 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), < 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.